CLINICAL TRIAL: NCT02778620
Title: Mean Systemic Filling Pressure and Heart Performance as Predictors of Successful Fluid Responsiveness in Patients With Aortic Valve Replacement
Brief Title: Mean Systemic Filling Pressure and Heart Performance Predicting Fluid Responsiveness in Aortic Valve Replacement
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, L.P.B. Meijs, MD, PhD-candidate Intensive Care Unit / resident cardiology, Catharina Ziekenhuis Eindhoven
Other Study IDs: M12-1270
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Cardiac Output, High
Keywords: Volume responsiveness mean systemic filling pressure
MeSH Terms: conditions — Cardiac Output, High

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aortic Valve Replacement: Post Anaesthetic Care Unit (PACU) patients treated with aortic valve replacement (AVR) are highly eligible for this study.These are patients with an indication for fast track treatment (PACU) post-cardiac surgery with a good left ventricular ejection fraction without significant co-morbidity. The final decision for PACU-classification is taken by the responsible anaesthesiologist and intensivist in close collaboration with the cardiothoracic surgeon performing the operation, as well as the cardiologist.

SUMMARY:
The purpose of this study is to determine fluid responsiveness in critically ill patients by measuring mean systemic filling pressure on the intensive care unit.

DETAILED DESCRIPTION:
The assessment of the cardiovascular state in critically ill patients is subject to difficulties in terms of the fact that several hemodynamic parameters, for example mean arterial blood pressure (MAP) and cardiac output (CO) supply insufficient information about the circulating volume and cardiac performance. There is a clinical need to adequate determination of intravascular volume status and therefore reliable predictors of fluid responsiveness are highly relevant. However, in determining the fluid status of a patient, the lack of appreciation of the venous side of the circulation persists today, which is greatly due to the inability to appropriately assess the venous side of the circulation. The importance of the venous part of the circulation is moreover reflected by the fact that an increase in venous resistance does reduce CO many times more than a similar increase in arterial resistance. Mean systemic filling pressure (Pms), which is defined as the pressure equal to the pressure which would be measured if the heart should suddenly stop pumping and all (arterial and venous) the pressures in the entire circulatory system should be brought to equilibrium instantaneously, is a good, complete and reliable reflection of the total intravascular fluid compartment. Passive leg raising (PLR) represents a "self-volume challenge" that predicts preload responsiveness and the transient hemodynamic changes on venous return can be directly monitored in ventilated patients, provided that there is an intact circulation, in order to test the amount of volume responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be older than 18 years, and must be equipped with a pulse-contour cardiac output system with a central venous catheter.
* Patients will be subsequently connected to the hemodynamic monitoring device Navigator™.
* In those patients with clinical signs of inadequate tissue perfusion, passive leg raising and standardized fluid challenge will be performed.

Exclusion Criteria:

* Patients with assist devices (e.g. intra aortic balloon pump, Impella®, ECMO), patients with arrhythmias (either atrial of ventricular) will be excluded from the study.
* Also, patients with inguinal impairment or contraindications for a passive leg raising will be excluded (such as deep venous thrombosis or elastic compression stocking), head trauma, an increase intra-abdominal pressure suspected by clinical context and examination as well as patients with absolute contraindications for fluid challenge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-aortic valve replacement patients
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2013-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Mean systemic filling pressure (Pms) | 1 hour
  An increase in mean systemic filling pressure after (self)volume-challenge indicating volume responsiveness of the patient

SECONDARY OUTCOMES:
Heart performance (eH) | 1 hour
  Quotient of driving pressure of venous return in mmHg

OTHER OUTCOMES:
Heart Rate | 1 hour
  Heart Rate in bpm
MAP | 1 hour
  Mean Arterial Blood Pressure
CI | 1 hour
  Cardiac Index
CVP | 1 hour
  Central Venous Pressure
SVR | 1 hour
  Systemic Vascular Resistance
PPV | 1 hour
  Pulse Pressure Variation
PVPI | 1 hour
  Pulmonary Vascular Permeability Index
pO2 | 1 hour
  Plethysmographic Oxygen Saturation
DO2I | 1 hour
  Delivery of Oxygen Index
Ventilation | 1 hour
  Mechanical Ventilation Settings
etCO2 | 1 hour
  End-tidal CO2
Temp perif | 1 hour
  Peripheral Temperature

CONTACTS AND LOCATIONS:
Overall Officials: Jan Bakker, MD, PhD, Study Chair — Erasmus Medical Center
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No
No, data remain anonymized within hospital and property of PI.